CLINICAL TRIAL: NCT04892706
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Vehicle Controlled, Clinical Study to Compare the Safety and Efficacy of IDP-126 Gel to Epiduo® Forte Gel (0.3% Adapalene/2.5% BPO), in the Treatment of Acne Vulgaris
Brief Title: Study to Compare the Safety and Efficacy of IDP-126 Gel to Epiduo® Forte Gel and Vehicle Gel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V01-126A-202
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IDP-126 Gel (Experimental): IDP-126 Gel (clindamycin phosphate 1.2%, BPO 3.1%, and adapalene 0.15%), applied topically to the face once daily for 12 weeks
  Interventions: Drug: IDP-126 Gel
- IDP-126 Vehicle Gel (Placebo Comparator): IDP-126 Vehicle Gel applied once daily for 12 weeks
  Interventions: Drug: IDP-126 Vehicle Gel
- Epiduo® Forte Gel (Active Comparator): Epiduo® Forte Gel (adapalene 0.3%/ 2.5% BPO) applied once daily for 12 weeks
  Interventions: Drug: Epiduo® Forte Gel

INTERVENTIONS:
Drug: IDP-126 Gel — Gel applied to face once daily in the evening.
  Other Names: IDP-126
  Arms: IDP-126 Gel
Drug: IDP-126 Vehicle Gel — Gel applied to face once daily in the evening.
  Other Names: Vehicle
  Arms: IDP-126 Vehicle Gel
Drug: Epiduo® Forte Gel — Gel applied to face once daily in the evening.
  Other Names: Epiduo® Forte
  Arms: Epiduo® Forte Gel

SUMMARY:
The safety and efficacy of once daily application of IDP 126 Gel will be compared to Epiduo® Forte and IDP-126 Vehicle Gel.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, vehicle-controlled, 12-week study designed to assess the safety, tolerability, and efficacy of IDP-126 Gel in comparison with Epiduo® Forte gel and IDP-126 Vehicle Gel at Weeks 2, 4, 8, and 12. To be eligible for the study, subjects must be at least 12 years of age and have a clinical diagnosis of moderate to severe acne (defined as an Evaluator's Global Severity Score [EGSS] of 3 or 4), presenting with 30-100 inflammatory facial lesions (papules, pustules, and nodules), 35-150 non-inflammatory facial lesions (open and closed comedones), and ≤ 2 facial nodules.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 12 years of age and older.
* Written and verbal informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit).
* Subject must have an EGSS of 3 (moderate) or 4 (severe) at the baseline visit.
* Subjects with a facial acne inflammatory lesion (papules, pustules, and nodules) count no less than 30, but no more than 100.
* Subjects with a facial acne non-inflammatory lesion (open and closed comedones) count no less than 35, but no more than 150.
* Subjects with 2 or fewer facial nodules.

Exclusion Criteria:

* Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gram negative folliculitis, dermatitis, eczema.
* Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
* Subjects with more than 2 facial nodules.
* Female subjects who are pregnant, nursing mothers, planning a pregnancy during the course of the study, or become pregnant during the study.
* Use of estrogens (eg, Depogen, Depo-Testadiol, Gynogen, Valergen, etc) for less than 12 weeks immediately preceding study entry; subjects treated with estrogens 12 or more consecutive weeks immediately prior to study entry need not be excluded unless the subject expects to change dose, drug or discontinue estrogen use during the study.
* Treatment of any type of cancer within the last 6 months, with the exception of complete surgical excision of skin cancer outside the treatment area.
* Subjects who have not undergone specified washout period(s) for topical preparations/physical treatments used on the face or subjects who require the concurrent use in the treatment area.
* Subjects who have not undergone specified washout period(s) for systemic medications or subjects who require the concurrent use of systemic medications.
* Subjects with any underlying disease that the investigator deems uncontrolled, and poses a concern for the subject's safety while participating in the study.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 686 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Study Director — Bausch Health Americas, Inc.
Locations (42):
- United States (34):
  - Bausch Site 134, Bryant, Arkansas
  - Bausch Site 118, Rogers, Arkansas
  - Bausch Site 110, Fremont, California
  - Bausch Site 101, Manhattan Beach, California
  - Bausch Site 106, San Diego, California
  - Bausch Site 112, San Diego, California
  - Bausch Site 128, San Diego, California
  - Bausch Site 105, Boynton Beach, Florida
  - Bausch Site 126, Clearwater, Florida
  - Bausch Site 135, North Miami Beach, Florida
  - Bausch Site 143, Sanford, Florida
  - Bausch Site 102, Tampa, Florida
  - Bausch Site 104, West Palm Beach, Florida
  - Bausch Site 122, West Palm Beach, Florida
  - Bausch Site 124, Newnan, Georgia
  - Bausch Site 127, Boise, Idaho
  - Bausch Site 129, Louisville, Kentucky
  - Bausch Site 139, Mandeville, Louisiana
  - Bausch Site 121, Metairie, Louisiana
  - Bausch Site 116, Rockville, Maryland
  - Bausch Site 103, Brighton, Massachusetts
  - Bausch Site 120, New Brighton, Minnesota
  - Bausch Site 108, Las Vegas, Nevada
  - Bausch Site 119, New York, New York
  - Bausch Site 133, New York, New York
  - Bausch Site 142, High Point, North Carolina
  - Bausch Site 109, Dublin, Ohio
  - Bausch Site 117, Oklahoma City, Oklahoma
  - Bausch Site 107, Gresham, Oregon
  - Bausch Site 114, Nashville, Tennessee
  - Bausch Site 111, Austin, Texas
  - Bausch Site 132, Houston, Texas
  - Bausch Site 123, Pflugerville, Texas
  - Bausch Site 137, Spokane, Washington
- Belgium (2):
  - Bausch Site 136, Kortrijk
  - Bausch Site 140, Maldegem
- Canada (6):
  - Bausch Site 138, Winnipeg, Manitoba
  - Bausch Site 125, Markham, Ontario
  - Bausch Site 141, Oakville, Ontario
  - Bausch Site 115, Peterborough, Ontario
  - Bausch Site 130, Waterloo, Ontario
  - Bausch Site 113, Saint-Jérôme, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gold M, Lain T, Harper JC, Baldwin H, Guenin E, Stein Gold L. Efficacy and Safety of Clindamycin Phosphate 1.2%/Adapalene 0.15%/Benzoyl Peroxide 3.1% Gel: Post Hoc Analysis by Baseline Disease Severity. Dermatol Ther (Heidelb). 2025 Jul;15(7):1867-1882. doi: 10.1007/s13555-025-01440-z. Epub 2025 May 16. PMID 40377868

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel | Epiduo® Forte Gel
Started | 230 | 228 | 228
Completed | 201 | 196 | 182
Not Completed | 29 | 32 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel | Epiduo® Forte Gel | Total
Number analyzed (Participants) | 230 | 228 | 226 | 684
Age, Continuous [Median (Full Range); unit: years] | 17.5 [12 to 56] | 17 [12 to 51] | 18 [12 to 51] | 17 [12 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 131 | 135 | 406
  Male | 90 | 97 | 91 | 278
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 0 | 3
  Asian | 16 | 27 | 19 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 24 | 28 | 26 | 78
  White | 179 | 160 | 165 | 504
  More than one race | 7 | 4 | 11 | 22
  Unknown or Not Reported | 4 | 6 | 5 | 15
Baseline Evaluator's Global Severity Score [Count of Participants; unit: Participants]
  Moderate | 201 | 204 | 198 | 603
  Severe | 29 | 24 | 28 | 81

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline to Week 12 in Lesion Counts.
Description: Inflammatory and non-inflammatory lesion counts were collected starting from the Baseline Visit.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Deviation); unit: lesion counts
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel | Epiduo® Forte Gel
Number analyzed (Participants) | 230 | 228 | 226
lesion counts | -29.9 (11.43) | -19.7 (13.11) | -27.9 (12.16)

2. Primary Outcome: Percentage of Subjects Who Achieve at Least a Two-grade Reduction From Baseline and Are "Clear" or "Almost Clear" at Week 12 in the Evaluator's Global Severity Score.
Description: The Evaluator's Global Severity Score has grades for acne severity of 0 (Clear), 1 (Almost Clear), 2 (Mild), 3 (Moderate), and 4 (Severe), with higher scores indicating worse severity.
Time Frame: Baseline to Week 12
Measure: Number; unit: participants
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel | Epiduo® Forte Gel
Number analyzed (Participants) | 230 | 228 | 226
participants | 118 | 41 | 74

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | IDP-126 Gel | IDP-126 Vehicle Gel | Epiduo® Forte Gel
All-Cause Mortality (participants affected / at risk) | 0/230 | 0/228 | 0/226
Serious Adverse Events (participants affected / at risk) | 1/230 | 0/228 | 0/226
Other Adverse Events (participants affected / at risk) | 23/230 | 0/228 | 16/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDP-126 Gel (N=230) | IDP-126 Vehicle Gel (N=228) | Epiduo® Forte Gel (N=226)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDP-126 Gel (N=230) | IDP-126 Vehicle Gel (N=228) | Epiduo® Forte Gel (N=226)
Application Site Pain (General disorders) | 23 (23) | 0 (0) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor for additional details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT04892706/Prot_SAP_000.pdf